CLINICAL TRIAL: NCT07336186
Title: The Impact of Virtual Reality-Assisted Relaxation on Breastfeeding Self-Efficacy and Breast Milk Production in Mothers of Premature Infants: A Randomized Controlled Trial
Brief Title: The Effect of Virtual Reality-Based Relaxation on Breast Milk Volume and Breastfeeding Self-Efficacy in Mothers of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Suzi Özdemir, Assistant Professor, PhD, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Suzi-04
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Lactation; Breastfeeding; Premature Birth; Maternal Stress; Self-Efficacy
Keywords: Virtual Reality; Relaxation techniques; Breast milk volume; Breastfeeding self-efficacy
MeSH Terms: conditions — Breast Feeding; Premature Birth

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either an experimental group receiving VR-based relaxation or a control group receiving standard care. Both groups were followed simultaneously for a period of three days to compare outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Mothers in this group used a virtual reality (VR) headset before the milk expression process. They watched a 10-minute relaxation video consisting of nature scenes (forests, waterfalls) accompanied by classical music. After the session, the researcher performed manual milk expression for at least 20 minutes. This procedure was repeated once daily for three days.
  Interventions: Behavioral: Virtual Reality-Based Relaxation
- Control Group (No Intervention): Mothers in this group received standard care. They sat in the same breastfeeding room for 10 minutes but did not use the VR headset or any other relaxation intervention. Following this period, the researcher performed manual milk expression for at least 20 minutes using the same technique as the experimental group. This procedure was repeated once daily for three days.

INTERVENTIONS:
Behavioral: Virtual Reality-Based Relaxation — A 10-minute immersive VR experience featuring calming nature landscapes and classical music designed to reduce stress and promote let-down reflex before milk expression.
  Arms: Virtual Reality Group

SUMMARY:
This study evaluates whether using virtual reality (VR) for relaxation helps mothers of premature babies produce more breast milk and feel more confident about breastfeeding. Mothers in the intervention group used VR headsets to watch calming nature videos while listening to music before expressing milk. The study compares their milk volume and self-efficacy scores to a control group receiving standard care.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact of a virtual reality (VR) relaxation intervention on breast milk production and breastfeeding confidence in mothers of premature infants.

Methodology:

* The study followed a randomized controlled design with two parallel groups.
* A total of 44 mothers whose infants were hospitalized in a Level II Neonatal Intensive Care Unit were enrolled.
* Participants were randomly assigned to either the intervention group or the control group.

Intervention and Procedures:

* Intervention Group: Participants used a VR headset to watch a 10-minute video featuring nature landscapes accompanied by classical music. Following the video, the researcher performed manual milk expression for at least 20 minutes.
* Control Group: Participants sat in the same breastfeeding room but did not use the VR headset. They received the same manual milk expression procedure by the same researcher.
* The procedure was conducted once daily for three consecutive days for both groups.
* To maintain stability in milk fat content, all sessions took place between 12:00 and 14:00.

Data Collection:

* Daily milk volume was measured in milliliters using sterile containers or injectors.
* Breastfeeding self-efficacy was assessed at the end of the third day using the "Breastfeeding Self-Efficacy Scale for Mothers of Preterm Infants".
* Demographic information was collected at the beginning of the study using a personal information form.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who have given birth to a single infant between 32 and 35 weeks of gestation.
* Mothers whose infants are hospitalized in the Neonatal Intensive Care Unit (NICU).
* Mothers who have delivered via Cesarean section.
* First-time mothers (Primiparous).
* Mothers who are willing to provide breast milk and participate in the study.
* Mothers whose infants are not yet able to breastfeed directly and require milk expression.

Exclusion Criteria:

* Mothers with any systemic or psychiatric diseases.
* Mothers with obstetric complications.
* Mothers who have a history of using addictive substances.
* Mothers who use medications or herbal products to increase breast milk (galactagogues).
* Mothers with hearing or vision impairments that would prevent the use of a VR headset.
* Mothers whose infants have congenital anomalies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Daily Breast Milk Volume | Daily for 3 consecutive days.
  The total amount of breast milk expressed manually during the study session.

SECONDARY OUTCOMES:
Breastfeeding Self-Efficacy Scale Score | At the end of the 3rd day of the intervention.
  Maternal confidence in breastfeeding as measured by the "Breastfeeding Self-Efficacy Scale for Mothers of Preterm Infants" (BSES-SF-PI). The scale consists of 20 items. Total scores range from 20 to 100, where higher scores indicate higher levels of breastfeeding self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT07336186/Prot_SAP_000.pdf